CLINICAL TRIAL: NCT06083025
Title: Influence of CleaRing Open-capsule Device on Refractive Predictability in Cataract Patients (Part 2)
Acronym: CleaRing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanita Lenses (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-0719 Part 2
Record Dates: First submitted 2023-10-05; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Posterior Capsule Opacification
Keywords: Posterior capsule opacification; Cataract; Ring
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single group, single center, open label study. Each study subject will be implanted bilaterally with IOL of surgeon's choice (same IOL in both eyes) and CleaRing device in one eye.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CleaRing device for cataract patients (Experimental): All subjects who meet eligibility requirements will be asked to participate. Subjects will be considered enrolled into the study after:
  1. A signed Informed Consent has been obtained.
  2. The subject has met all of the inclusion and none of the exclusion criteria.
  3. The ability of the subject to safely undergo cataract surgery under local anesthesia was confirmed by the investigator, according to standard procedure of the medical center.
  Interventions: Device: CleaRing

INTERVENTIONS:
Device: CleaRing — The Hanita CleaRing device is an intraocular implant designed for inhibition of PCO leading to reduction in the Nd:YAG treatment rate. The device is implanted into the capsular bag after the extraction of the crystalline lens and prior to implantation of the IOL. The device is manufactured by Hanita Lenses from a hydrophilic acrylic co-polymer which is being used for the production of Intra-ocular lenses.

SUMMARY:
The Hanita CleaRing device is an intraocular implant designed for inhibition of PCO leading to reduction in the Nd:YAG treatment rate. The device is implanted into the capsular bag after the extraction of the crystalline lens and prior to implantation of the IOL. The device is manufactured by Hanita Lenses from a hydrophilic acrylic co-polymer which is being used for the production of Intra-ocular lenses.

DETAILED DESCRIPTION:
Cataract surgery has undergone significant improvement in terms of surgical technique, instrumentation and the quality of intraocular lenses (IOLs) over the past decades. Although the rate of posterior capsular opacification (PCO) has decreased, it is still the most common complication following uneventful cataract surgery, with the rate of laser capsulotomy ranging from 10% to 37%1-5 ND:YAG capsulotomy is a highly successful treatment, but it is not free of complications, such as increased intraocular pressure (IOP), pitting or dislocation of the IOL, cystoid macular edema, and retinal detachment. PCO also places an economic burden on the healthcare system. The importance of PCO prevention has increased in recent years, due to the expanding popularity of premium IOLs. Patients implanted with a premium IOL usually have high demands with regard to outcome, and PCO can also have an earlier effect on the performance of a premium IOL (i.e., multifocal IOLs).

Previous attempts to prevent PCO have included investigations of various IOL materials and designs, surgical techniques, and pharmacological materials. Unexpectedly lower PCO rates were recently noticed in eyes that were implanted with a special type of IOL, e.g., the Synchrony IOL (AMO, Santa Ana, CA, USA)8 and the FluidVision IOL (PowerVision, Belmont, CA, USA). It was hypothesized that the capsular bag stayed open due to the special design of these IOLs, and that this should reduce the PCO rate. Based upon this concept, a special open capsule ring was designed for intracapsular implantation in an attempt to maintain the capsular bag open and to reduce PCO rate. Safety and efficacy of the device was demonstrated through several animal studies. The tested devices were effective in reducing posterior capsule opacification and Soemmering's ring formation by 69% to 77% compared to control group. The Hanita CleaRing device is designed to be implanted in the capsular bag together with a standard posterior chamber IOL in a minimally invasive cataract surgery. The device is intended to reduce posterior capsular opacification leading to reduced Nd:YAG treatment rate. The raw material of the device is a hydrophilic co-polymer, considered to be biocompatible and practically inert to the eye tissue. The objective of this study is to evaluate the safety and the efficacy of CleaRing device in cataract patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 50 and 80 years of age
* Subject is designated for bilateral cataract surgery
* Both eyes fulfil the following criteria:

  * Potentially able to achieve a good vision (by opinion of the investigator)
  * ACD is at least 2.5mm (from epithelium)
  * Corneal astigmatism is at most 2.0 dpt
  * Axial length is between 22.0 and 26.0 mm
  * Able to obtain pupil dilation of at least 6.0 mm
  * Average keratometry values between 42.0 and 46.0 D
* Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed

Exclusion Criteria:

* Subject diagnosed with glaucoma of any type or having intraocular pressure above 24mmHg
* Subject who has undergone previous intraocular surgery
* Subject with corneal abnormality that would prevent stable and reliable refraction
* Subject with weak or torn zonules
* Subject with Pseudoexfoliation syndrome (PEX)
* Subject with amblyopia
* Subject with retinal disease that in the opinion of the principal investigator would prevent stable and reliable refraction or might be worsened due to implantation of the device
* Subject is diagnosed with active anterior segment intraocular inflammation
* Subject is obligated to previous participation in another study with any investigational drug or device within the past 30 days
* Subject is pregnant

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The first primary objective of this study is to evaluate the influence of Clearing open-capsule device on refractive predictability in cataract patients. | 1, 3 and 5 years
  Refractive will be evaluated by Automated refraction
The second primary objective of this study is to evaluate the influence of Clearing open-capsule device on refractive predictability in cataract patients. | 1, 3 and 5 years
  Refractive will be evaluated by subjective refraction
The third primary objective of this study is to evaluate the influence of Clearing open-capsule device on refractive predictability in cataract patients. | 1, 3 and 5 years
  Refractive will be evaluated by visual acuity measurement.

SECONDARY OUTCOMES:
Secondary objective of this study is to evaluate the influence of the device on PCO rate | 1, 3 and 5 years
  PCO will be evaluated by using Biomicroscopy (Slit Lamp)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Kleinmann, Prof., Principal Investigator — Wolfson MC
Locations (1):
- Wolfson Medical Center, Holon, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No